CLINICAL TRIAL: NCT02647710
Title: PHAT Life: Preventing HIV/AIDS Among Teens in Juvenile Justice
Acronym: PHAT Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Geri Donenberg, Associate Dean of Research, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MD005861 (NIH); 5R01MD005861-05 (NIH)
Record Dates: First submitted 2015-12-29; First posted 2016-01-06 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: HIV
Keywords: HIV Prevention; Juvenile Justice; Sexual Health; Evidence Based Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PHAT Life Intervention (Experimental): PHAT Life: Preventing HIV/AIDS Among Teens, is a uniquely-tailored intervention designed for recently-arrested juvenile offenders on probation. The program will teach teens about HIV/AIDS, sexually transmitted infections, and safer decision-making. PHAT Life draws on social learning theory and a Social-Personal Framework to address individual and social mechanisms related to HIV-risk, including emotion regulation, peer norms, partner communication, relationship characteristics, and HIV/AIDS/STI and substance use knowledge, attitudes, and beliefs.
  Interventions: Behavioral: PHAT Life Intervention
- Health Promotion Control (Active Comparator): A health promotion program focusing on nutrition, physical activity, substance use, and sexual health.
  Interventions: Behavioral: Health Promotion Control

INTERVENTIONS:
Behavioral: PHAT Life Intervention — HIV Prevention behavioral health intervention
  Arms: PHAT Life Intervention
Behavioral: Health Promotion Control — Behavioral health intervention control
  Arms: Health Promotion Control

SUMMARY:
PHAT Life: Preventing HIV/AIDS Among Teens, is a uniquely-tailored intervention designed for recently-arrested juvenile offenders on probation. The program will teach teens about HIV/AIDS, sexually transmitted infections, and safer decision-making. The PHAT Life Research Study is a 2-arm randomized controlled trial of the PHAT Life Intervention. The investigators will test and compare PHAT Life to the health promotion control group on adolescent risky sexual behavior, substance use, and theoretical mediators.

DETAILED DESCRIPTION:
High rates of mental illness, HIV/AIDS/STI, and incarceration among African Americans (AA) reflect significant health disparities, particularly among youth. Teens in juvenile justice are disproportionately AA, and compared to the general population, juvenile offenders (JO) report more risky sexual behavior, drug and alcohol use, and psychiatric disorders, and are more likely to test positive for STIs. Still, few empirically-supported, theoretically-driven programs exist to address their negative health outcomes. This proposal addresses these health disparities by testing an innovative and uniquely tailored HIV/AIDS/STI, mental health, and substance use program designed for and pilot tested with recently arrested 13 - 17 year-old urban males and females (85% African American, 14% Latino/a) released on probation. PHAT Life was derived from a carefully staged process that included an active, diverse, multi-disciplinary advisory board, a youth advisory board, focus groups, two pilot tests, extensive feedback, and a series of curriculum revisions over three years. The R34 established feasibility and acceptability, revealed positive youth and stakeholder feedback, and yielded good preliminary outcomes at 3-month follow-up (e.g., increased condom use) to justify an efficacy trial. This application proposes a 2-arm randomized controlled trial to test PHAT Life versus a health promotion program with recently arrested 13-17 year-old male and female, mostly ethnic minority JO (as representative of Cook County) on probation in Chicago. The investigators will use the procedures and methods established in the developmental study to recruit, enroll, assess, track, and intervene with teens. Investigators will randomly assign youth to PHAT Life (N=150) or a health promotion control group (N=150). The interventions will be delivered in single sex groups of 5 - 7 teens at Evening Reporting Centers. Assessments will occur at baseline, 6-, and 12-months post-treatment, and participants will be screened for three common STIs (Chlamydia, Gonorrhea, Trichamonas) at baseline and 12-month follow-up. All youth who test positive for an STI will receive single dose antibiotic treatment free of charge. An intent-to-treat analysis will be used to test and compare PHAT Life to the health promotion control group on adolescent risky sexual behavior, substance use, and theoretical mediators. This study answers a compelling need for innovative prevention programs that address the intersecting health disparities of mental illness and HIV/AIDS/STIs among youth in juvenile justice. Without intervention, these teens continue to engage in risk behaviors post-release, amplifying their own and their partner's risk for HIV/AIDS/STIs. The lasting effects on community well-being, individual employment prospects, and neighborhood health are profound, but effective programs can alter the negative developmental trajectories of this very high-risk population and begin to redress existing health disparities.

ELIGIBILITY:
Inclusion Criteria:

* male or female gender
* placed on probation following arrest
* remanded to a probation program
* 13-17 years old
* both adolescent and parent are fluent English speakers
* not a ward of the state (DCFS Ward).

Exclusion Criteria:

* are unable to understand the consent/assent process
* do not speak English, because instruments are normed for English speakers
* do not assent; d) legal guardians do not consent to teens' participation
* are not 13 -17 years old
* are not on probation or remanded to a probation program
* are Wards of the state (DCFS Ward)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 349 (Actual)
Dates: Start 2010-06-15 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in HIV/STI Risk Behaviors at 6 and 12 months | baseline, 6-months, and 12--months
  AIDS Risk Behavior Assessment (ARBA) A computer-assisted structured interview of self-reported sexual behavior and drug use derived from five well-established measures. The outcomes include ever had sex, condom use, number of partners, sex while using drugs and/or alcohol.

SECONDARY OUTCOMES:
Change in HIV/AIDS/STI Knowledge, Attitudes, Beliefs, and Behavioral Skills at 6 and 12 months | Baseline, 6-months, and 12-months
  Survey measuring knowledge regarding transmission routes, misconceptions about transmission, and risk-reduction strategies; attitudes and beliefs including peer norms, intentions to prevent HIV/AIDS/STI, attitudes towards preventive actions, and beliefs about condom use; as well as self-efficacy to prevent transmission, apply condoms, and negotiate with a partner.
Change in mental health symptoms at 6 and 12 months | Baseline, 6-months, and 12-months
  The Youth Self Report (YSR) is a widely-used and validated measure of child behavior problems that generates raw and T-scores for internalizing and externalizing syndromes as well as narrow-band problems (e.g., delinquency, anxiety, depression).
Change in Partner Sexual Communication at 6 and 12 months | Baseline, 6-months, and 12-months
  Questionnaire in which participants indicate whether they ever talked to their romantic or dating partners and sexual partners about a list of sexual topics, how often they discussed them, and whether they talk was open and comfortable. Items were adapted from the Sexual Risk Behavior Questionnaire.
Change in Relationship dynamics at 6 and 12 months | Baseline, 6-months, and 12-months
  The Sexual Relationship Power Scale (SRPS) measures perceptions of relationship control and decision-making dominance. It has good internal consistency and predictive and constructed validity.
Change in trauma symptoms and violence exposure at 6 and 12 months | Baseline, 6-months, and 12-months
  The UCLA PTSD Index will measure exposure to trauma and violence.
Change in peer influences at 6 and 12 months | Baseline, 6-months, and 12-months
  The Peer Convention Behavior Questionnaire will measure peer support of risky behavior, peer norms, and peer pressure and teens' association with prosocial peers.
Change in parental Influences at 6 and 12 months | Baseline, 6-months, and 12-months
  The Parenting Style Questionnaire (PSQ) measures parental supervision, monitoring, and permissiveness.
Change in parental communication at 6 and 12 months | Baseline, 6-months, and 12-months
  The Parent-Child Sexual Communication Questionnaire assesses youths' perceived quality and quantity of risk-specific communication with their parents.
Biological Measure of N. Gonorrhoeae Acquisition | 12-months
  Sexually transmitted infections will be measured using biological endpoint (yes/no) to evaluate intervention effects. Participants will be screened for N. gonorrhoeae and treated if necessary at baseline. They will be tested again 12 months later to determine rate of STI acquisition.
Biological Measure of C. Trachomatis Acquisition | 12-months
  Sexually transmitted infections will be measured using biological endpoint (yes/no) to evaluate intervention effects. Participants will be screened for C. trachomatis and treated if necessary at baseline. They will be tested again 12 months later to determine rate of STI acquisition.
Biological Measure of T. Vaginalis Acquisition | 12-months
  Sexually transmitted infections will be measured using biological endpoint (yes/no) to evaluate intervention effects. Participants will be screened for T. vaginalis and treated if necessary at baseline. They will be tested again 12 months later to determine rate of STI acquisition.

CONTACTS AND LOCATIONS:
Overall Officials: Geri Donenberg, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Donenberg GR, Emerson E, Mackesy-Amiti ME, Udell W. HIV-Risk Reduction with Juvenile Offenders on Probation. J Child Fam Stud. 2015 Jun 1;24(6):1672-1684. doi: 10.1007/s10826-014-9970-z. PMID 26097376
- [Background] Udell W, Donenberg G, Emerson E. Parents matter in HIV-risk among probation youth. J Fam Psychol. 2011 Oct;25(5):785-9. doi: 10.1037/a0024987. PMID 21875199
- [Background] Wilson HW, Berent E, Donenberg GR, Emerson EM, Rodriguez EM, Sandesara A. Trauma History and PTSD Symptoms in Juvenile Offenders on Probation. Vict Offender. 2013;8(4):10.1080/15564886.2013.835296. doi: 10.1080/15564886.2013.835296. PMID 24273468
- [Result] Donenberg G, Emerson E, Kendall AD. HIV-risk reduction intervention for juvenile offenders on probation: The PHAT Life group randomized controlled trial. Health Psychol. 2018 Apr;37(4):364-374. doi: 10.1037/hea0000582. Epub 2018 Feb 1. PMID 29389155
- [Result] Kendall AD, Emerson EM, Hartmann WE, Zinbarg RE, Donenberg GR. A Two-Week Psychosocial Intervention Reduces Future Aggression and Incarceration in Clinically Aggressive Juvenile Offenders. J Am Acad Child Adolesc Psychiatry. 2017 Dec;56(12):1053-1061. doi: 10.1016/j.jaac.2017.09.424. Epub 2017 Oct 5. PMID 29173739